CLINICAL TRIAL: NCT01012128
Title: Comparison of Temporal Artery, Axillary, and Rectal Temperatures in Preterm Infants in the NICU
Brief Title: Comparison of Three Methods of Taking Temperatures in the Newborn Intensive Care Unit
Status: Withdrawn | Type: Observational
Why Stopped: Closed: logistical problems that could not be resolved.
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Michael F. Bruno, MD, Christiana Care Health System
Other Study IDs: 600687
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Thermometry
Keywords: Temporal Artery Thermometer; Temperature; Preterm Infants

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Preterm infants will have their body temperature measured by three different devices in order to evaluate whether the newest device, a temporal artery scanning thermometer, is accurate for patients in the preterm period.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants corrected to 30-35 weeks gestation
* current incubator set on air control between 28-30 degrees centigrade

Exclusion Criteria:

* infants <30 and >35 weeks gestation
* infants requiring > 30 degrees centigrade in incubator on air control
* infants currently not in an incubator

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infants corrected to 30-35 weeks gestation
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of temporal artery thermometer measurements | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Bruno, MD, Principal Investigator — Christiana Hospital / Christiana Care Health System
Locations (1):
- Christiana Hospital, Newark, Delaware, United States